CLINICAL TRIAL: NCT01742637
Title: A Multi-Center, Double-Blind, Randomized, Placebo Controlled, Parallel-Group Study Comparing Adapalene and Benzoyl Peroxide Gel 0.1%/2.5% (Taro Pharmaceuticals Inc.) to Epiduo® (Galderma Laboratories, L.P., Adapalene and Benzoyl Peroxide Gel 0.1%/2.5%) and Both Active Treatments to a Placebo in the Treatment of Acne Vulgaris.
Brief Title: Study Comparing Adapalene and Benzoyl Peroxide Gel 0.1%/2.5% to Epiduo® and Both to a Placebo Control in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADBG-1206, 1302
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Adapalene and Benzoyl Peroxide Gel 0.1%/2.5%; Epiduo®
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adapalene and Benzoyl Peroxide Gel 0.1%/2.5% (Experimental): Adapalene and Benzoyl Peroxide Gel 0.1%/2.5% (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Adapalene and Benzoyl Peroxide Gel 0.1%/2.5%
- Epiduo® Gel (Active Comparator): Epiduo® (Adapalene and Benzoyl Peroxide Gel 0.1%/2.5%) (Galderma Laboratories, L.P.)
  Interventions: Drug: Epiduo® Gel
- Placebo (Placebo Comparator): Placebo (vehicle of test product) (Taro Pharmaceuticals Inc.)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adapalene and Benzoyl Peroxide Gel 0.1%/2.5% — Adapalene and Benzoyl Peroxide Gel 0.1%/2.5% (Taro Pharmaceuticals Inc.)applied topically once daily for 84 consecutive days.
  Arms: Adapalene and Benzoyl Peroxide Gel 0.1%/2.5%
Drug: Epiduo® Gel — Epiduo® (Adapalene and Benzoyl Peroxide Gel 0.1%/2.5%) (Galderma Laboratories, L.P.)applied topically once daily for 84 consecutive days.
  Arms: Epiduo® Gel
Drug: Placebo — Placebo (vehicle of test product) (Taro Pharmaceuticals Inc.)applied topically once daily for 84 consecutive days.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the therapeutic equivalence and safety of Adapalene and Benzoyl Peroxide 0.1%/2.5% Gel (Taro Pharmaceuticals Inc.) and Epiduo® (Adapalene and Benzoyl Peroxide 0.1%/2.5% Gel) (Galderma Laboratories, L.P.) in the treatment of acne vulgaris, and to demonstrate the superiority of the efficacy of the test and reference products over the vehicle (placebo) control in the treatment of acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non pregnant female aged ≥ 12 and ≤ 40 years with a clinical diagnosis of acne vulgaris.
* Subjects who are 18 years of age or older must have provided written informed consent. Subjects 12 to 17 years of age must have provided written assent, which must be accompanied by written informed consent from the subject's legally acceptable representative. All subjects or their legally acceptable representatives must sign a Health Insurance Portability and Accountability Act authorization.
* Subjects must have a minimum of ≥ 25 non-inflammatory lesions and ≥ 20 inflammatory lesions and ≤ 2 nodulocystic lesions, at baseline on the face.
* Subjects must have a definite clinical diagnosis of acne vulgaris severity grade 2, 3, or 4 as per the Investigator's Global Assessment (IGA).
* Subjects must be willing to refrain from using all other topical acne medications or antibiotics for acne vulgaris during the 12-week treatment period, other than the investigational product.
* Female subjects of childbearing potential (excluding those who are surgically sterilized or postmenopausal for at least 1 year), in addition to having a negative urine pregnancy test, must be willing to use an acceptable form of birth control during the study from the day of the first dose administration to 30 days after the last administration of study drug.
* All male subjects must agree to use accepted methods of birth control with their partners, from the day of the first dose administration to 30 days after the last administration of study drug.
* Subjects must be willing and able to understand and comply with the requirements of the protocol.
* Subjects must be in good health and free from any clinically significant disease, including but not limited to, conditions that may interfere with the evaluation of acne vulgaris.
* Subjects who use make-up must have used the same brands/types for a minimum period of 14 days prior to study entry and must agree to not change brand/type or frequency of use throughout the study.

Exclusion Criteria:

* Female subjects who are pregnant, nursing or planning to become pregnant during study participation.
* Subjects with a history of hypersensitivity or allergy to adapalene, retinoids and/or any of the study medication ingredients, have a known hypersensitivity to adapalene and benzoyl peroxide and its excipients.
* Subjects with the presence of any skin condition that would interfere with the diagnosis or assessment of acne vulgaris.
* Subjects with excessive facial hair that would interfere with diagnosis or assessment of acne vulgaris.
* Subjects who have performed wax depilation of the face within 14 days prior to baseline.
* Subjects who have used within 6 months prior to baseline or use during the study of oral retinoids or therapeutic Vitamin A supplements of greater than 10,000 units/day.
* Subjects who have used estrogens or oral contraceptives for less than 3 months prior to baseline.
* Subjects who have used any of the following procedures on the face within 1 month prior to baseline or use during the study: cryodestruction or chemodestruction, dermabrasion, photodynamic therapy, acne surgery, intralesional steroids, x-ray therapy.
* Subjects who have used any of the following treatments within 1 month prior to baseline or use during the study: systemic steroids, systemic antibiotics, systemic treatment for acne vulgaris, systemic anti-inflammatory agents.
* Subjects who have used any of the following treatments within 2 weeks prior to baseline or during the study: topical steroids, topical retinoids, α-hydroxy/glycolic acid, benzoyl peroxide, topical anti-inflammatory agents, topical antibiotics.
* Use of spironolactone is prohibited during the study.
* Use of tanning booths, sunbathing, or excessive exposure to the sun are prohibited during the study.
* Subjects who have received radiation therapy and/or anti-neoplastic agents within 90 days prior to baseline.
* Subjects who have unstable medical disorders that are clinically significant or have life-threatening diseases.
* Subjects who have on-going malignancies requiring systemic treatment, and subjects who have any malignancy of the skin of the facial area.
* Subjects who engage in activities that involve excessive or prolonged exposure to sunlight or weather extremes, such as wind or cold.
* Subjects who consume excessive amounts of alcohol or use drugs of abuse.
* Subjects who have participated in an investigational drug study within 30 days prior to baseline.
* Subjects who have been previously enrolled in this study.
* Subjects who have had laser therapy, electrodesiccation and phototherapy to the facial area within 180 days prior to study entry.
* Subjects who have had cosmetic procedures which may affect the efficacy and safety profile of the investigational product within 14 days prior to study entry. Cosmetic procedures and facials are prohibited throughout the study.
* Subjects who currently have or have recently had bacterial folliculitis on the face.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2008 (Actual)
Dates: Start 2012-10; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Inflammatory and non-inflammatory lesion counts | Week 12
  Percent change from baseline to week 12 in the inflammatory (papules and pustules) and non-inflammatory (open and closed comedones) lesion counts.

SECONDARY OUTCOMES:
Clinical response of success. | Week 12
  The proportion of subjects with a clinical response (IGA) of success at week 12. Success should be defined as an IGA score that is at least 2 grades less than the baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Catawba Research, Study Chair — http://catawbaresearch.com/contact/